CLINICAL TRIAL: NCT00803127
Title: VS-Sense Result Reading Clarity
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Collaborators: Lin Medical Center, Haifa (Other); Common Sense (Other)
Responsible Party: hadar kessary, common sense
Other Study IDs: F-7-25.2-1
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Vaginitis
Keywords: vaginal infection, color appearance
MeSH Terms: conditions — Vaginitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — VAGINAL DISCHARGE

GROUPS / COHORTS (1):
- no treament
  Interventions: Device: vs-sense

INTERVENTIONS:
Device: vs-sense — detection swab

SUMMARY:
This study is designed to demonstrate the result reading clarity of the VS-SENSE is substantially equivalent to the result reading clarity of the Nitrazine pH Paper test for vaginal secretions.

DETAILED DESCRIPTION:
Once informed consent has been signed, the clinician will perform the following:

Record baseline variables in the CRF. The 1st clinician will obtain a vaginal secretion sample by using the VS-SENSE swab. The 1st clinician will obtain the specimen by separating the labia to expose the vagina. The yellow tip of the VS-SENSE swab will be inserted into the vagina approximately 5 cm/ 2". The 1st clinician will use the VS-SENSE according the instructions for use - attachment 1 to the protocol.

The 1st clinician will read the VS-SENSE results and record them on the designated form (Clinician Report - VS-SENSE Result form), and fill out the table regarding the VS-SENSE reading clarity on the same form.Vaginal examination (including speculum examination) - will be performed by a 2nd clinician, masked from the results of the 1st clinician test.

The 2nd clinician will use a vaginal swab for pH measurement by Nitrazine pH Paper test. The Nitrazine pH Paper test will be performed according to strict manufacturer's instruction.

The 2nd clinician will read the results of the Nitrazine pH Paper test result, document it on the Clinician Report - pH Test Result form, and fill out the table regarding the pH test reading clarity on the same form.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic women, ages 18 and above.
2. Subjects willing and able to sign the informed consent form.

Exclusion Criteria:

1. Subjects are unable or unwilling to cooperate with study procedures.
2. Subjects are currently participating in other clinical study that may directly or indirectly affect the results of this study.
3. Women with blood present in their vaginal secretion.
4. Subjects that have had sexual relations or applied vaginal douched within the previous 12 hours.
5. Subjects that applied vaginal medications within the last 3 days.
6. Subjects with symptoms and signs of pelvic inflammatory disease.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Symptomatic and asymptomatic women, ages 18 and above.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
The clinician reports of the VS-SENSE test results, the pH measurement by Nitrazine Paper test records, and the results reading clarity grade from the clinician. | 5 minuts

CONTACTS AND LOCATIONS:
Locations (1):
- Lin Medical center, Haifa, West Galil, Israel